CLINICAL TRIAL: NCT05556629
Title: Quantitative Testing of Patient and Healthcare Provider Knowledge, Attitudes, and Behavior About NATPARA® (Parathyroid Hormone) for Injection, for Subcutaneous Use
Brief Title: A Survey to Assess Participants' and Physicians' Knowledge, Attitudes and Behavior When Using NATPARA
Acronym: NATPARA KAB
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: TAK-834-4008; EUPAS48713 (Registry Identifier: ENCePP (EU PAS))
Record Dates: First submitted 2022-09-23; First posted 2022-09-27 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Hypoparathyroidism
MeSH Terms: conditions — Hypoparathyroidism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- NATPARA: Participants: Participants who have been approved for NATPARA and a part of the special use program (SUP) prior to survey implementation will participate in the survey via telephone or internet.
  Interventions: Other: No Intervention
- NATPARA: Healthcare Provider (Prescribing Physician): Healthcare provider (HCPs)/Prescribing physician who can provide a 10-digit National Provider Identifier (NPI) number and who are certified in the NATPARA risk evaluation and mitigation strategy (REMS) by successfully completing the NATPARA REMS program training module for prescribing physicians, including the knowledge assessment, and submitting a NATPARA REMS Program Prescriber Enrollment Form will participate in the survey via telephone or internet.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
This main aim of this study is to check the level of knowledge and assess attitudes and behaviors of both participants and prescribing physicians regarding the risks and safe use of NATPARA. The survey will be done via internet, telephone, or paper and participants will be able to choose the method that is preferred. No study medicines will be provided to patients in this study.

ELIGIBILITY:
Participant inclusion criteria:

• Participants who are 18 years of age or older and who have been approved for NATPARA and a part of the SUP Program prior to survey implementation are eligible to participate in the survey.

* A caregiver may participate in this survey on behalf of a participant who is a part of the SUP Program and who is eligible but unable to complete the survey.

Prescribing physician inclusion criteria:

• HCPs in the United States (US) who can provide a 10-digit NPI number and who are certified in the NATPARA REMS by successfully completing the NATPARA REMS Program Training Module for Prescribing Physicians, including the Knowledge Assessment, and submitting a NATPARA REMS Program Prescribing Physician Enrollment Form are eligible for participation in the survey and a part of the SUP Program.

Participant and Prescribing Physician exclusion criteria:

* Respondents who do not agree to participate in the survey will be excluded.
* Survey respondents who have been employed or whose immediate family members have been employed by NPS, Shire, Takeda, United BioSource LLC, (UBC), or the Food and Drug Administration (FDA) are not eligible to participate in the survey and will be excluded.
* Respondents who reported having a conflict of interest will be excluded.
* Respondents who are not part of the SUP program will be excluded.

Participant exclusion criteria:

* Participants who do not agree to participate in the survey will be excluded.
* Participants who have opted out of receiving communications will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who have been approved for NATPARA and a part of the SUP program prior to survey implementation and prescribing physicians who can provide a 10-digit NPI number and who are certified in the NATPARA REMS by successfully completing the NATPARA REMS program training module for prescribing physicians, including the knowledge assessment, and submitting a NATPARA REMS program prescribing physician enrollment form are eligible for participation in the survey.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants and Prescribing Physicians Providing Correct Responses to Questions | Up to approximately 7 years
  All question for key risk message and about NATPARA will be asked through a questionnaire, Participant or prescribing physicians (HCPs) would need to respond true or false to each question based upon understanding and knowledge. Respondents could be participants or HCPs.

SECONDARY OUTCOMES:
Number of Participants and Prescribing Physicians Providing At Least 80 Percent (%) Correct Responses to Each key Risk Messages | Up to approximately 7 years
  The questions will be asked to participants and HCPs will be counted as correct if 80% of the correct responses are provided and not more than one incorrect response is provided. In key risk message, general question about NATPARA will be asked, participant or HCPs would need to respond true or false to each question based upon understanding and knowledge. Respondents could be participants or HCPs.
Number of Participants and Prescribing Physicians who Demonstrated Understanding of Each key Risk Messages | Up to approximately 7 years
  Understanding demonstration is defined as respondents who answered 80% or more questions/items in a key risk message correctly. In key risk message, general question about NATPARA will be asked, participants or HCPs would need to respond true or false to each question based upon understanding and knowledge. Respondents could be participants or HCPs.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (1):
- Shire-NPS Pharmaceuticals, INC. (Shire now part of Takeda), Lexington, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/7e4fd13264a44033?idFilter=%5B%22TAK-834-4008%22%5D